CLINICAL TRIAL: NCT00785382
Title: A Randomized, Placebo Controlled Trial of Pregabalin for Postoperative Pain in Women Undergoing Breast Cancer Surgery
Brief Title: Pregabalin for Postoperative Pain in Women Undergoing Breast Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant Professor, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IWK-4298-2008
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Postoperative Pain
Keywords: Pain, Pregabalin, Lyrica, Breast surgery
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Pregabalin 150 mg

INTERVENTIONS:
Drug: Placebo — Lactulose Placebo
  Arms: 1
Drug: Pregabalin 150 mg — 150 mg Q12H x 2 doses
  Other Names: Lyrica
  Arms: 2

SUMMARY:
We hypothesize that pregabalin will decrease postoperative pain, as measured by the surrogate markers postoperative pain rating scores and postoperative opioid consumption while improving the quality of recovery following breast cancer surgery compared to placebo. The primary outcome will be postoperative pain, measured by a NRS and the quality of recovery score (QoR) in the first 24h postoperative period. Do women undergoing breast cancer surgery with general anesthesia and receiving pregabalin prior to their surgery and 12 hours later have lower NRS and a greater QoR score in the first 24 hours after their surgery than those women who received placebo?

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesia physical status class I & II
2. Age ¬< 65 years
3. English-speaking
4. Unilateral breast cancer surgery without axillary node dissection (i.e. simple mastectomies and lumpectomies +/- "sentinal" node biopsy)

Exclusion Criteria:

1. Known or suspected allergy, sensitivity, or contraindication to pregabalin
2. Known or suspected allergy to morphine, NSAIDs, acetaminophen or oxycodone
3. Morbid Obesity (Body Mass Index ≥ 45 kg/m2)
4. History of a seizure disorder
5. Pregnancy
6. Current pre-operative therapy with pregabalin, gabapentin, or any opioid
7. Any other physical or psychiatric condition which may impair their ability to cooperate with postoperative study data collection
8. CrCl < 60 ml/min [CrCl = 0.85 x ((140 - age) x weight(kg)) / (72 x Cr(mg/dL)))]

Max Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be postoperative pain, measured by a NRS and the quality of recovery score (QoR) in the first 24h postoperative period. | 24 hours

SECONDARY OUTCOMES:
NRS / QoR - 48 hour Opioid Consumption Side effects - nausea, sedation | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD FRCPC, Principal Investigator — IWK
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada